CLINICAL TRIAL: NCT05092880
Title: Radioembolization in Elderly/Fragile Patients With Unresectable Livermetastases of Colorectal Cancer, CAIRO7 Study of the DCCG
Brief Title: Radioembolization in Elderly/ Fragile Patients With mCRC
Acronym: CAIRO7
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Dutch Colorectal Cancer Group (Other)
Responsible Party: Principal Investigator, Marnix G.E.H. Lam, MD, PhD, Professor of Nuclear Medicine, UMC Utrecht
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAIRO7
Record Dates: First submitted 2021-07-30; First posted 2021-10-26 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Colorectal Cancer Metastatic

STUDY DESIGN:
Intervention Model Description: randomized phase 2
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Standard of care first-line systemic therapy (Active Comparator): capecitabine plus anti-VEGF antibody
  Interventions: Drug: Standard of care first-line systemic therapy
- Radioembolization (Experimental): radioembolization of liver with holmium-166 microspheres
  Interventions: Device: radioembolization

INTERVENTIONS:
Device: radioembolization — holmium-166 microspheres
  Arms: Radioembolization
Drug: Standard of care first-line systemic therapy — Capecitabine plus anti-VEGF antibody
  Arms: Standard of care first-line systemic therapy

SUMMARY:
Radioembolization (RE) is a minimally invasive treatment with administration of radioactive microspheres into the hepatic artery via a microcatheter. Since tumors are preferentially supplied by the hepatic artery, most microspheres get trapped in the tumor. RE has been shown a feasible and safe procedure for the treatment of unresectable CRC liver metastases. These data compare favourably with the toxicity data of capecitabine plus bevacizumab, but this should be validated in a prospective study.

The proposed study investigates the efficacy of RE as an alternative, better tolerated and more cost-effective treatment option in elderly or frail patients compared to chronic systemic treatment with comparable progression-free survival.

DETAILED DESCRIPTION:
Rationale In The Netherlands, ±14.000 people/year are diagnosed with colorectal cancer (CRC), and 50% of patients already have/will develop distant metastases, most commonly to the liver. Standard treatment is palliative systemic treatment, which prolongs overall survival (OS). In only a small subset of patients with liver-only metastases, local treatment (i.e. surgery) of metastases is possible with curative intent, either initially or after downsizing by intensive systemic treatment. The average age at CRC diagnosis is 69 yrs, and 30% of CRC patients are ≥75 yrs. Thus, many patients are too old and/or fragile to allow intensive systemic regimens or major surgery. In frail/elderly patients the standard treatment is capecitabine plus an antibody against the vascular endothelial growth factor (VEGF, i.e. bevacizumab or biosimilar), given until disease progression or unacceptable toxicity, resulting in a median progression free survival (PFS) of 8.5-9.2 months. Capecitabine-induced hand-foot syndrome and diarrhoea are the most commonly occurring toxicities. Prolonged exposure to CTCAE grade 2 toxicity in frail or elderly patients may already significantly impact quality of life and daily functioning. Therefore, treatments with less toxicity would be of great value for these patients.

Radioembolization (RE) is a minimally invasive treatment with administration of radioactive microspheres into the hepatic artery via a microcatheter. Since tumors are preferentially supplied by the hepatic artery, most microspheres get trapped in the tumor. RE has been shown a feasible and safe procedure for the treatment of unresectable CRC liver metastases. These data compare favourably with the toxicity data of capecitabine plus bevacizumab, but this should be validated in a prospective study.

The proposed study investigates the efficacy of RE as an alternative, better tolerated and more cost-effective treatment option in elderly or frail patients compared to chronic systemic treatment with comparable progression-free survival.

Objectives:

Primary objective:

The objective of this randomized phase 2 study is to demonstrate efficacy of a single RE in terms of PFS in CRC patients with liver-only metastases who are candidates for palliative systemic treatment with capecitabine plus anti-VEGF antibody (bevacizumab or biosimilar).

Secondary objectives:

* To evaluate safety/toxicity.
* To evaluate cost-effectiveness.
* To evaluate quality of life (QoL).
* To evaluate overall survival.

Study design:

Multi-center, interventional, treatment, randomized phase 2, open label, comparative study. The study will be conducted within the network of the Dutch Colorectal Cancer Group (DCCG). Patients will be randomized 1:1 between RE and systemic treatment with capecitabine + anti-VEGF antibody.

Study population:

220 elderly and/or fragile patients with liver-limited, unresectable metastatic colorectal cancer, previously not systemically treated, who are candidates for systemic treatment with capecitabine plus an anti-VEGF antibody, will be enrolled in this study. Given the lack of validated selection criteria for elderly and/or frail this judgement will be left to the discretion of the local investigator.

Intervention:

Individualized holmium-166 radioembolization (166Ho-RE) will be performed via a catheter during angiography. Dosimetry-based treatment planning will be individualized using Q-Suite™ software. The comparator, standard systemic treatment, will be given by the local investigator and will consist of capecitabine orally 1000 mg/m2 bid day 1-14 + anti-VEGF antibody i.v. 7.5 mg/kg day 1 at 3-weekly cycles, continued until disease progression or unacceptable toxicity.

Main study parameters/endpoints:

Primary endpoint:

Progression-free survival.

Secondary endpoints:

* Safety/toxicity.
* Cost-effectiveness.
* QoL.
* Overall survival.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have given written informed consent.
2. Female or male patients aged ≥18 years.
3. Metastatic colorectal cancer, with metastases confined to the liver, previously not systemically treated.
4. Previous local treatment of liver metastases by resection of a maximum of two liver segments and/or local ablation is allowed.
5. Elderly/frail patients, according to the local investigator not eligible for local treatments or intensive systemic regimens with combination chemotherapy.
6. ECOG Performance status 0-2 (Table 1).
7. Eligible for systemic treatment with capecitabine + anti-VEGF antibody.
8. Adequate bone marrow (Hb ≥ 6 mmol/L, WBC ≥ 3x109/L, platelets ≥ 100x109/L), liver (serum bilirubin ≤ 1x upper limit of normal (ULN), ASAT/ALAT ≤ 5x ULN), and renal (GFR ≥ 40 ml/min) functions.

Exclusion Criteria:

1. Previous systemic treatment for metastatic disease.
2. Previous adjuvant treatment completed within 6 months prior to randomization.
3. Symptoms of primary tumour, if in situ, that require intervention; prior treatment with (chemo)radiotherapy and/or resection of primary tumor is allowed.
4. Resection of more than 2 liver segments, 2-stage procedures and/or radiotherapy of liver metastases.
5. Eligible for more intensive systemic regimens (i.e. doublet or triplet chemotherapy).
6. Eligible for local treatment of liver metastases (e.g. surgical resection, ablation).
7. Presence of extrahepatic metastases; the presence of small (≤ 1 cm) lesions outside the liver on CT scan that are not clearly suspicious for metastases and/or the presence of enlarged hilar lymph nodes in the liver up to a maximal diameter of 2 cm is allowed.
8. Non-correctable INR >2.0.
9. Any serious comorbidity preventing the safe administration of anti-VEGF antibody treatment. This includes uncontrolled hypertension or treatment with ≥3 antihypertensive drugs, arterial (cerebro)vascular event within the past 12 months, history of bleeding, history of GI perforation, or presence of fistulae.
10. Pregnancy or breastfeeding.
11. Mental disorders that may compromise patient compliance.
12. Active second malignancy within the previous 5 years, with the exception of adequately treated basal cell carcinoma of skin and in situ carcinoma of cervix.
13. Body weight over 150 kg (because of maximum table load).
14. Known severe allergy for intravenous contrast fluids.
15. Participation to another investigational study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | 4 years

SECONDARY OUTCOMES:
Adverse event frequency and grade according to CTCAE version 5.0 | 3.5 years
Quality of life (EORTC quality of life questionnaire number C30) | 3.5 years
  For all questionnaires the official manuals will be used to calculate the subscales.
Quality of life (EORTC quality of life questionnaire number CR29) | 3.5 years
  For all questionnaires the official manuals will be used to calculate the subscales.
Quality of life (Multidimensional Fatigue Inventory: MFI-20) | 3.5 years
  For all questionnaires the official manuals will be used to calculate the subscales.
Overall survival | 5 years
Cost-effectiveness: Medical Consumption Questionnaire (MCQ) | 4 years
  For all questionnaires the official manuals will be used to calculate the subscales.
Cost-effectiveness: Productivity Cost Questionnaire (PCQ) | 4 years
  For all questionnaires the official manuals will be used to calculate the subscales.

CONTACTS AND LOCATIONS:
Locations (1):
- UMC Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No